CLINICAL TRIAL: NCT00250016
Title: 1102C-T. Pharmacology Study of Aerosolized Liposomal-Nitro-20 (S)-Camptothecin (L9NC) in Patients With Metastatic or Recurrent Cancer of the Endometrium. Tissue Submission for Patients With Endometrial Cancer.
Brief Title: Pharmacology Study of Aerosolized Liposomal 9-Nitro-20 (S)-Camptothecin (L9NC)
Status: Withdrawn | Type: Observational
Why Stopped: UNM did not proceed with research
Sponsor: University of New Mexico (Other)
Responsible Party: Claire F. Verschraegen, M.D.; Principal Investigator, University Of New Mexico - CRTC
Other Study IDs: 1102C-T
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Corpus Uteri; Endometrial Cancer
Keywords: Endometrium; Tissue; L9NC
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample, tumor endometrial tissue, and normal endometrial tissue.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine the amount of Aerosolized Liposomal-Nitro-20 (S)-Camptothecin (L9NC) in a patients blood and tumor.

DETAILED DESCRIPTION:
Patients on this study are being asked to allow the researchers to take a piece of some normal endometrial tissue and tumor tissue. No additional endometrial tissue will be taken for this study other than what is surgically indicated to resect the patients tumor completely. Prior to this surgery, patients will receive one more dose of L9NC in the outpatient clinic in the same manner as the other L9NC treatments they have received. After the tumor has been removed, the tissue will be examined by a pathologist, who will take what is needed to diagnose the residual disease. What is not needed for patient care will be used for research. A piece of the tumor and some normal endometrial tissue surrounding the tumor will be sent to the Investigational Drug Program laboratory, which is located in the Cancer Center, to measure the amount of drug that is left in the patients tumor. The patients tissue will be kept until all tissues are collected from all patients, which could take up to 10 years. The tissue will not be used for any other purpose. The samples will be labeled with the patients initials.

ELIGIBILITY:
Inclusion Criteria:

* Patients participating in Phase II Study of Aerosolized Liposomal 9-Nitro-20 (S)- Camptothecin (L9NC) in Patients with Metastatic or Recurrent Cancer of the Endometrium are eligible.

Exclusion Criteria:

* Not specified.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients participating in the trial - "Phase II Study of Aerosolized Liposomal-Nitro-20 (S)-Camptothecin (L9NC) in Patients with Metastatic or Recurrent Cancer of the Endometrium"
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2003-08 (Actual); Primary Completion 2007-04 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claire F Verschraegen, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States